CLINICAL TRIAL: NCT04733118
Title: Chemotherapy-Free pCR-Guided Strategy With Subcutaneous Trastuzumab-pertuzumab and T-DM1 in HER2-positive Early Breast Cancer (PHERGAIN-2)
Brief Title: Chemotherapy-Free pCR-Guided Strategy With Trastuzumab-pertuzumab and T-DM1 in HER2-positive Early Breast Cancer
Acronym: PHERGAIN-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP293
Record Dates: First submitted 2020-12-04; First posted 2021-02-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient HER 2+ IHC 3+ (Experimental): Patients ≥18 years of age with previously untreated HER2-positive (HER2[+]) (Immunohistochemistry [IHC] 3+) invasive carcinoma according to the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) criteria and tumor size between >5 to 25 mm by breast magnetic resonance imaging (MRI) and node-negative status by clinical exam, MRI, and ultrasound. Patients must have not been previously treated with chemotherapy, anti-HER2 therapy, radiation therapy, or endocrine therapy (ET) for invasive breast cancer. Patients with metastatic disease are not eligible. In patients with suspected axillary node involvement, a negative fine needle aspiration biopsy (FNAB) will be mandatory
  Interventions: Drug: Trastuzumab and Pertuzumab (FDC SC) and T-DM1

INTERVENTIONS:
Drug: Trastuzumab and Pertuzumab (FDC SC) and T-DM1 — Patients will receive Trastuzumab and Pertuzumab as a subcutaneous fixed-dose combination (PH FDC SC) (± ET depending on HR status) for 8 3-week cycles, on day 1 only. ET will consist of letrozole for post-menopausal women or tamoxifen ± ovarian function suppression (OFS) for pre-menopausal women administered continuously. Men will receive tamoxifen.
  After completing neoadjuvant therapy, a final breast MRI will be performed 2 weeks prior to surgery. Surgery will be performed within 4 weeks after completion of the last cycle of PH FDC SC.
  Adjuvant systemic therapy will start within 4 weeks from surgery. There will be three different cohorts depending on pathological report:
  * Cohort A: PH FDC SC ± ET for 10 additional 3-week cycles
  * Cohort B: T-DM1 ± ET for 10 cycles
  * Cohort C: T-DM1 ± ET for 10 cycles, with possibility of physician's choice chemotherapy before adjuvant T-DM1.
  Other Names: Trastuzumab emtansine; Phesgo; Kadcyla

SUMMARY:
This is a multicenter, open-label, single-arm, one-stage, phase II study to assess the efficacy of a chemotherapy-free pathological complete response (pCR)-guided strategy with trastuzumab and pertuzumab (given as a subcutaneous fixed-dose combination) and T-DM1, for patients with previously untreated HER2-positive early breast cancer.

DETAILED DESCRIPTION:
Patients ≥ 18 years of age with previously untreated HER2 IHC 3+ invasive carcinoma according to ASCO/CAP 2018 guidelines.

Tumor size between >5 to 30 mm by breast MRI and node-negative status by clinical exam, MRI, and ultrasound. In patients with suspected axillary node involvement, a negative fine needle aspiration biopsy (FNAB) will be mandatory.

Central review for:

Breast MRI. HER2 status. Neoadjuvant treatment will consist In 8 cycles of fixed-dose subcutaneous (SC FDC) HP combination (± ET according to HR status).

urgery will be performed within 4 weeks from the last cycle of HP (sentinel node biopsy will be mandatory; subsequent axillary dissection will be performed according to local guidelines). Surgery will require free margins for any infiltrating or DCIS lesion.

Radiotherapy will be mandatory for patients with breast preservation.

Adjuvant systemic therapy will be started within 4 weeks from surgery depending on pathological report:

Arm A: pCR (breast and axilla): HP SC FDC x 10 cycles. Arm B: Residual invasive breast tumor and/or ypN0(i+), ypN0(mol+), ypN1mi: T-DM1 x 10 cycles Arm C: ypN1 to N3: T-DM1 x 10 cycles, with physician's choice chemotherapy allowed between surgery and T-DM1.

All patients with HR[+] tumors will receive adjuvant ET up to at least 5 years (ET will also be administered in association with adjuvant HP or T-DM1, with the exception of the cycles involving the use of chemotherapy in Arm C).

ELIGIBILITY:
Inclusion criteria

Patients will be included in the study only if they meet ALL of the following criteria:

1. Written informed consent prior to beginning specific protocol procedures.
2. Female or male patients ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically proven invasive carcinoma of the breast.
5. Tumor size must be between ≥ 5mm and ≤30mm in greatest dimension using breast MRI. Note: Although tumors between ≥ 5mm and ≤ 10mm are not considered target lesions by RECIST v1.1, we will consider these lesions as targets to follow-up.
6. Patients must have node-negative breast cancer by clinical exam, MRI and ultrasound according to the American Joint Committee on Cancer (AJCC) 8th edition.
7. Centrally confirmed HER2[+] status with IHC score 3+.
8. Known estrogen receptor (ER) and progesterone receptor (PgR) status prior to study entry that should be performed by immunohistochemical methods according to the local institution standard protocol.
9. Patients with multifocal or multicentric breast cancer are eligible; patients with 2 lesions or less are eligible only if both lesions are sampled and meet the inclusion criteria #5, #6, and #7.
10. Normal left ventricular function and diastolic function (left ventricular ejection fraction [LVEF] ≥55%) as assessed by echocardiogram or multiple-gated acquisition scan (MUGA) documented within ≤28 days prior to first dose of study treatment.
11. Adequate bone marrow, liver, and renal function:

    1. Hematological: White blood cell (WBC) count > 3.0 × 109/L, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100.0 × 109/L, and hemoglobin ≥ 10.0 g/dL (≥ 6.2 mmol/L).
    2. Hepatic: total bilirubin ≤ institutional upper limit of normal (ULN) (except for Gilbert's syndrome); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 times ULN.
    3. Renal: serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
    4. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
12. Patient must be accessible for treatment and follow-up.
13. Willingness and ability to provide blood samples at baseline, C3D1 before treatment infusion, pre-surgery and then after surgery: every 6 months for the first 5 years, and every year thereafter until the EoS.
14. Willingness and ability to provide tumor tissue samples at baseline and at surgery.
15. Women of childbearing potential and men with partners of childbearing potential must be willing to use one highly effective form of nonhormonal contraception or two effective forms of nonhormonal contraception by the patient and/or partner and to continue its use for the duration of study treatment and for seven months after the last dose of study treatment.

    Note: Acceptable forms of effective contraception should include two of the following:

    i. Placement of non-hormonal intrauterine device (IUD) ii. Condom with spermicidal foam/gel/film/cream/suppository iii. Diaphragm or cervical/vault caps with spermicidal foam/film/cream/suppository The above contraception is not a requirement in the case the male patient, or male partner of a female patient, is surgically sterilized, the female patient is post-menopausal or the patient remains abstinent and truly abstains from sexual activity (refrains from heterosexual intercourse).
16. Negative serum pregnancy test for premenopausal women including women who have had a tubal ligation and for women less than 12 months after the onset of menopause.

Exclusion criteria:

Any patient meeting ANY of the following criteria will be excluded from the study:

1. Any previous treatment, including chemotherapy, anti-HER2 therapy, radiation therapy, or ET for invasive breast cancer (except for breast carcinoma in situ of the contralateral breast cancer, in the last five years before treatment initiation in this study).
2. HER2 disease with IHC score 0, 1+ or 2+ and in situ hybridization (ISH) positive result.
3. Evidence of metastatic disease. Note: All patients must be willing to undergo chest and pelvis computed tomography (CT)/MRI scan before enrolment to prove no evidence of metastatic disease. Bone scan will be performed at baseline only if there is suspicion of bone metastases. If a bone scan cannot be performed, an alternative is PET/CT using 18F-labeled sodium fluoride (18F-fluoride PET/CT).
4. Patients with bilateral breast cancer.
5. Known hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances.
6. History of other malignancy within the last five years prior to first dose of study drug administration, except for curatively treated basal and squamous cell carcinoma of the skin and/or in situ cervical carcinoma.
7. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) despite adequate antihypertensive treatment.
8. Serious cardiac illness or medical conditions including, but not confined to, the following:

   * History of NCI CTCAE v5.0 Grade ≥ 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) Class ≥ II.
   * High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate ≥ 100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block, such as second-degree AV-block Type 2 [Mobitz II] or third-degree AV-block).
   * Serious cardiac arrhythmia or severe conduction abnormality not controlled by adequate medication.
   * Angina pectoris requiring anti-angina medication.
   * Clinically significant valvular heart disease.
   * Evidence of transmural infarction on electrocardiogram (ECG).
   * Evidence of myocardial infarction within the last 12 months prior to study entry.
9. History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction [LVSD], left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome.
10. Active uncontrolled infection at the time of enrollment.
11. Current known infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
12. Patients with pulmonary disease requiring continuous oxygen therapy.
13. Grade ≥2 neuropathy as per National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v)5.0.
14. Previous history of bleeding diathesis.
15. Patient is currently receiving chronic treatment with corticosteroids, or another immunosuppressive agent (standard premedication for chemotherapy and local applications are allowed).
16. Major surgical procedure or significant traumatic injury within 14 days prior to study entry or anticipation of need for major surgery within the course of the study treatment.
17. Any other concurrent severe and/or uncontrolled medical condition that would contraindicate patient participation in the clinical study.
18. History of having received any investigational treatment within 28 days prior to study entry.
19. Pregnant or breast-feeding women or patients not willing to apply highly effective contraception as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
3-year recurrence-free interval (3y-RFI) | 3 years
  3-year recurrence-free interval (3y-RFI) defined as time from start of treatment in adjuvant setting until recurrence, new invasive disease, or death from breast cancer. Recurrence will be defined in accordance with the standardized efficacy endpoints (STEEP) criteria.
Global health status decline | 1 year
  Global health status decline rate at 1 year from start of neoadjuvant treatment, defined as the rate of patients with a ≥10% global health status decline at 1 year from start of neoadjuvant treatment as assessed by the Global Health Status/QoL EORTC-QLC-C30 scale and its breast cancer module QLQ-BR23.

SECONDARY OUTCOMES:
pathological complete response (pCR) | after neoadjuvant treatment (8 cycles, an average of 6months)
  pCR rates concerning breast and lymph nodes (pCRBREAST+LYMPH NODE) and pCR concerning breast only (pCRBREAST) in the overall population.
pathological complete response (pCR) according to hormone receptor (HR) status | after neoadjuvant treatment (8 cycles, an average of 6months)
  pCR rates according to HR status
Residual cancer burden (RCB) | after neoadjuvant treatment (8 cycles, an average of 6months)
  RCB -0, -I, -II, -III; (0:best outcome, III: worst outcome)
Breast-conserving surgery (BCS) | after neoadjuvant treatment (8 cycles, an average of 6months)
  Evaluate the rate of BCS
Response rate BCS | after neoadjuvant treatment (8 cycles, an average of 6months)
  Evaluate the correlation between final MRI-guide response rate results and breast-conserving surgery (BCS)
Response rate pCR | after neoadjuvant treatment (8 cycles, an average of 6months)
  Evaluate the correlation between final MRI- guide response rate and pCR
Response rate RCB | after neoadjuvant treatment (8 cycles, an average of 6months)
  Evaluate the correlation between final MRI -guide response rate and RCB at surgery
Survival rates EFS | 3 years and 5 years
  Analyze the event-free survival (EFS)
Survival rates relapse-free survival (RFS) | 3 years and 5 years
  Analyze RFS
Survival rates invasive disease-free survival (iDFS) | 3 years and 5 years
  Analyze iDFS
Survival ratesdistant relapse-free survival (DRFS) | 3 years and 5 years
  Analyze DRFS
Survival rates disease-free survival (DFS) | 3 years and 5 years
  Analyze DFS
Survival rates overall survival (OS) | 3 years and 5 years
  Analyze OS
Survival ratesbreast cancer-specific survival (BCSS). | 3 years and 5 years
  Analyze BCSS
Survival rates relapse-free interval (RFI) | 5 years
  Analyze RFI
Safety adverse events (AEs) | Baseline up to 3 years
  Number of patients with treatment-related AEs (Grade 3 and 4 AEs and serious adverse events [SAEs]) by using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
Safety adverse events (AEs) | Baseline up to 5 years
  Number of patients with treatment-related AEs (Grade 3 and 4 AEs and serious adverse events [SAEs]) by using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
Health-Related Quality of Life (HRQoL) - QLQ-C30 | Baseline up to 5 years
  Change from baseline in scores using the European Organisation for Research and Treatment of Cancer QoL Questionnaire Core 30 (QLQ-C30) [with 5 functional and 3 symptom scales, a Global Health Status (GHS)/QoL scale, and 6 single items], at baseline, Day 1 of cycles 2-4, then on Day 1 of each subsequent cycle starting with cycle 6, and at the end-of-treatment. Responses to all items are converted to a 0-100 scale using a standard scoring algorithm. For functional scales, higher score represents a better level of functioning; for symptom scales, a higher score represents a higher severity of symptoms.
Health-Related Quality of Life (HRQoL) - QLQ-BR23 | Baseline up to 5 years
  Change from baseline in scores using the European Organisation for Research and Treatment of Cancer QLQ-BR23 [with 4 functional and 4 symptom scales], at baseline, Day 1 of cycles 2-4, then on Day 1 of each subsequent cycle starting with cycle 6, and at the end-of-treatment. Responses to all items are converted to a 0-100 scale using a standard scoring algorithm. For functional scales, higher score represents a better level of functioning; for symptom scales, a higher score represents a higher severity of symptoms.
To assess the cardiac toxicity profile after 1 year of adjuvant treatment | after 1 year of adjuvant treatment
  Adverse events of cardiotoxicity after 1 year of adjuvant treatment according to the NCI-CTCAE v.5.0.
To assess the general toxicity profile according to CTCAE v.5.0. | at 3 and 5 year
  Toxicity and safety profile at 3 and 5 years as per NCI-CTCAE v.5.0.
To evaluate the ratio of patients who have needed chemotherapy. | before T-DM1
  Ratio of patients of cohort C who will receive adjuvant chemotherapy before T-DM1.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart-Cussac, MD, Principal Investigator — Arnau de Vilanova Hospital, Valencia (Spain)
Locations (41):
- UMHAT Sveti Ivan Rilski EAD Department of Medical Oncology, Sofia, Bulgaria
- Germany (6):
  - Praxisnetzwerk Hämatologie und intern. Onkologie, Cologne
  - Evangelisches Krankenhaus Bethesda, Duisburg
  - Kliniken Essen Mitte, Essen
  - Universitätsklinikum Essen Frauenklinik, Essen
  - Universitätsklinikum Mannheim GmbH, Manheim
  - Klinikum Ernst von Bergmann, Potsdam
- Hungary (2):
  - Békés county hospital, Békés
  - Tolna County Balassa János Hospital, Szekszárd
- Italy (7):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - AO Ospedale Civile Legnano, Milan
  - Istituto Europeo di Oncologia - NC, Milan
  - Ospedale San Gerardo, Monza
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Spain (25):
  - ICO L'Hospitalet - Instituto Catalán de Oncología, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Universitari San Joan de Reus, Reus, Tarragona
  - Centro Oncológico de Galicia, A Coruña
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Institut Català d' Oncologia Badalona (ICO), Badalona
  - Hospital Universitari Dexeus - Grupo Quirónsalud, Barcelona
  - VHIO Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Consorcio Hospitalario Provincial De Castelló, Castellon
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Complejo Hospitalario de Jaen, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Quirón San Camilo- Ruber Juan Bravo, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario de Torrejón, Torrejón
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital La Fe, Valencia
  - Consorcio Hospital General de Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No